CLINICAL TRIAL: NCT06800755
Title: Evaluation of the Efficacy and Tolerance of the Medical Device RL3020-DP0364 in Adult Population With Stable Mild Plaque Psoriasis, Dry Skin and Pruritus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RL302020240210
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis; Pruritus; Dry Skin
Keywords: Psoriasis; Pruritus; Dry Skin; Medical Device
MeSH Terms: conditions — Psoriasis; Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults with stable mild plaque psoriasis, dry skin and pruritus (Experimental): Device: Dexeryl (RL3020-DP0364) Tested product is applied twice a day. The maximum duration of application is 30 days.
  Interventions: Device: Dexeryl (RL3020-DP0364)

INTERVENTIONS:
Device: Dexeryl (RL3020-DP0364) — Product application on body (head excluded)

SUMMARY:
The product RL3020-DP0364 developed by Pierre Fabre Laboratories moisturizes durably and repairs dry or atopic skin, especially in the case of certain dermatoses (atopic dermatitis, ichthyosis, etc ...) and erythema induced by radiotherapy. Its unique formula treats the symptoms of dry skin by creating a protective film that prevents dehydration and helps protect the skin from external aggressions.

Through this study, the efficacy of this medical device will be evaluated specifically in subjects presenting stable psoriasis, dry skin and pruritus with an application on the whole body (excluding the head).

ELIGIBILITY:
Inclusion criteria:

* Subject with stable mild plaque psoriasis covering ≤ 10% BSA (Body Surface Area; excluding the head*)
* Subject whose plaque psoriasis has been diagnosed for at least 6 months before the inclusion visit
* Subject with dry skin according to the investigator assessment
* Subject with a pruritus intensity (on average over the previous 24 hours) ≥ 3 on a Numerical Rating Scale (NRS) between 0 and 10 (with 0 = no pruritus and 10 = worst imaginable pruritus) on the body*

  * the head is not included in the evaluated area

Exclusion criteria:

Criteria related to the disease:

* Subject with erythrodermic psoriasis, pustular psoriasis
* Subject with palmoplantar keratoderma
* Subject with any other aetiology of pruritus, not related to plaque psoriasis
* Subject with history of allergy or intolerance to any of the tested product ingredients
* Subject having any other dermatologic condition than psoriasis, or characteristics (like tattoo, wound…) on body liable to interfere with the study assessments
* Subject having an acute, chronic or progressive disease or history of disease liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements

Criteria related to treatments and/or products:

* Biotherapy treatment in the 6 months prior to the inclusion visit or ongoing or planned to be started during the study
* Other systemic treatment for psoriasis (acitretin, cyclosporine, methotrexate, apremilast...) in the 3 months prior to the inclusion visit or ongoing or planned to be started during the study
* Phototherapy treatment in the 4 weeks prior to the inclusion visit or ongoing or planned to be started during the study
* Any other systemic treatment incompatible with the study or liable to interfere with the study assessments according to the investigator, in the weeks prior to the inclusion visit, ongoing or planned to be started during the study
* Topical treatment for psoriasis (corticosteroid, vitamin D analogs…) applied on the body* in the 4 weeks prior to the inclusion visit or ongoing or planned to be started during the study
* Topical product (including any moisturizer, emollient, keratolytic …) applied on the body* in the 7 days prior to the inclusion visit or ongoing or planned to be started during the study
* Any product applied on the body* before the visit, the day of inclusion visit
* Any other topical treatment or product applied on the body* incompatible with the study or liable to interfere with the study assessments according to the investigator, in the weeks prior to the inclusion visit, ongoing or planned to be started during the study

  * the head is not included in the evaluated area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-07-04 (Estimated); Study Completion 2025-07-04 (Estimated)

PRIMARY OUTCOMES:
Pruritus intensity assessment | 29±2 days
  The pruritus intensity on the whole body (head excluded) (on average over the previous 24 hours) will be assessed by the subject at Visit 1 (Day 1-before product application) and at Visit 3 (Day 29(±2)) according to the following [0-10] Numerical Rating Scale

SECONDARY OUTCOMES:
Average pruritus intensity assessment (previous 24hours) | Day 1, Day 8, Day 14±2, Day 29±2
  The pruritus intensity will be assessed on the whole body (head excluded), on average over the previous 24 hours by the subject, according to NRS (Numerical Rating Scale)
Average pruritus intensity assessment (previous 7 days) | Day 1, Day 8, Day 14±2, Day 29±2
  The pruritus intensity will be assessed on the whole body (head excluded), on average over the previous 7 days by the subject, according to NRS (Numerical Rating Scale)
Worst pruritus intensity assessment (previous 7 days) | Day 1, Day 8, Day 14±2, Day 29±2
  The worst pruritus intensity will be assessed on the whole body (head excluded), over the previous 7 days by the subject, according to NRS (Numerical Rating Scale)
Pruritus severity and impact on quality-of-life assessment | Day 1, Day 14±2, Day 29±2
  pruritus severity and impact on quality of life will be assessed by the subject with a Patient Reported Outcome (PRO) questionnaire including 20 questions
Pruritus characteristics assessment | Day 1, Day 29±2
  Pruritus characteristics (duration, degree, direction, disability and distribution) will be assessed by the subject with a global score (1 global score considering all characteristics) on the 5-D itch scale
mPASI assessment | Day 1, Day 14±2, Day 29±2
  mPASI (modified Psoriasis Area Severity Index) (excluding the head) will be assessed by the investigator on a scale ranged from 0 to 64,8
Xerosis intensity assessment | Day 1, Day 14±2, Day 29±2
  Xerosis intensity on the whole body outside psoriasis plaques and the xerosis intensity on psoriasis plaques will be assessed by the investigator using the following scale ranged from 0 to 4: 0= None, 1= Mild, 2= Moderate, 3= Severe, 4= Very severe
Tolerance assessment | Day 29±2
  Assessment of the tolerance by the investigator with the attribution of one of the 5 levels, considering all individual Adverse Events and their characteristics based on the following 5-point scale (excellent = 5 to bad = 0)
Acceptability questionnaire assessment | Day 29±2
  Acceptability questionnaire regarding the use of the product will be completed by the subject
Illustrative photographs assessment | Day 1, Day 14±2, Day 29±2
  Photographs of a representative area of psoriasis

CONTACTS AND LOCATIONS:
Locations (1):
- Dermscan Poland, Gdansk, Poland, Poland